CLINICAL TRIAL: NCT04030000
Title: A Pilot Phase II Trial of Intravenous Paclitaxel and Intraperitoneal Carboplatin/Taxol Followed by Radiation in Patients With Advanced Stage Uterine Serous Carcinoma
Brief Title: Uterine Serous Carcinoma and Adjuvant Combined Intraperitoneal Chemotherapy and Radiation
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: could not enroll anyone due to staff changes
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Karin Shih, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: USC
Record Dates: First submitted 2019-04-05; First posted 2019-07-23 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Uterine Carcinoma
MeSH Terms: interventions — CP protocol

STUDY DESIGN:
Intervention Model Description: During Week 1-18, subjects will be placed on open-label IP Carboplatin/IV Paclitaxel on Day 1, then administered IP Paclitaxel on Day 8. This will be repeated every 3 weeks for 6 cycles. A CT imaging scan will be performed after six cycles of chemotherapy, prior to radiation. Also, in Week 19-23, subjects will receive Pelvic radiation therapy (IMRT) if deemed necessary. Additionally, from Week 24-26, High Dose Radiation or IMRT will be used where appropriate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Paclitaxel/Carboplatin and radiation (Other): Paclitaxel 135 mg/m2 over 3 hrs on day 1 Carboplatin IP (AUC= 6.0) on day 1 Paclitaxel 60 mg/m2 IP on Day 8 Repeat q 21 days x 6 cycles
  Pelvic 6MV Photon Beam Energy, or IMRT where appropriate 1.8 Gy Dose/FX Total Dose 45 Gy
  High Dose Radiation (HDR) x 3, or IMRT where appropriate 5 Gy to 0.5cm Depth from the Vaginal Cylinder Surface Total Dose 15 Gy
  Interventions: Drug: Paclitaxel/Carboplatin; Radiation: Pelvic radiation therapy

INTERVENTIONS:
Drug: Paclitaxel/Carboplatin — IV paclitaxel in combination with IP carboplatin
Radiation: Pelvic radiation therapy — EBRT and vaginal brachytherapy

SUMMARY:
Uterine serous carcinoma (USC) is an uncommon, but aggressive variant of endometrial carcinoma that has poor response to standard therapy. After staging and surgery, radiation therapy and/or chemotherapy is recommended to treat patients at high risk for recurrence. In advanced stage and recurrent setting, high risk uterine cancer mirrors ovarian cancer with it spread patterns and response to therapy. Based on these findings and the similarities as well as the clinical success of paclitaxel with IP platinum therapy in patients with ovarian serous carcinoma, investigators propose to prospectively assess IV/IP therapy in patients with advanced stage and recurrent USC.

During Week 1-18, subjects will be placed on open-label IP Carboplatin/IV Paclitaxel on Day 1, then administered IP Paclitaxel on Day 8. This will be repeated every 3 weeks for 6 cycles. A CT imaging scan will be performed after six cycles of chemotherapy, prior to radiation. Also, in Week 19-23, subjects will receive Pelvic radiation therapy (IMRT) if deemed necessary. Additionally, from Week 24-26, High Dose Radiation or IMRT will be used where appropriate.

Patients will be monitored for toxicity and feasibility of the regimen. Secondary outcomes will include assessing the frequency and the reasons for early discontinuation of the study treatments as well as describing patient-reported quality of life parameters at specified time points during the study using validated questionnaires: EORTC QLQ-C30 and QLQ-OV28.

DETAILED DESCRIPTION:
TREATMENT PLAN 5.1 Dosing Guidelines 5.1.1 Chemotherapy Paclitaxel is available commercially. Paclitaxel 135mg/m2 will be given over 1 hour in 250-500 ml of 5% dextrose or normal saline. Premedication for prevention of anaphylactic reactions with anti-histamines and/or steroids should be administered as per standard practice. Paclitaxel should be given first given the risk of immediate drug sensitivity reaction. Following on Day 8 of the cycle, paclitaxel will be given IP at 60mg/m2. After infusion the patient will be asked to change position at 15-minute intervals for two hours to ensure adequate intra-abdominal distribution. No attempt will be made to retrieve the infusate, however if a large amount of ascites is present, ascites may be drained by paracentesis or accessed port prior to instillation of drug.

Carboplatin is available commercially. Carboplatin should be reconstituted in 500-1000cc of normal saline warmed to 37 °C (when feasible) and infused through a peritoneal catheter as rapidly as possible. It is preferred that an additional 1000 ml of warm saline is infused after IP Carboplatin, or 500ml of warmed normal saline infused before and after IP Carboplatin to help with drug dispersion throughout the peritoneal cavity, for a total volume of approximately two liters. After infusion the patient will be asked to change position at 15-minute intervals for two hours to ensure adequate intra-abdominal distribution. No attempt will be made to retrieve the infusate, however if a large amount of ascites is present, ascites may be drained by paracentesis or accessed port prior to instillation of drug. Carboplatin at an AUC of 6.0 will be administered intraperitoneally (if there is a prior history of radiotherapy, AUC of 5 would be used). AUC based dosing as described by Calvert et al. will be according to the following formula: Dose (mg) = AUC x (GFR + 25).

The initial GOG trial using combination paclitaxel and carboplatin therapy was performed on patients with optimally debulked ovarian epithelial carcinoma.40 At that time, the carboplatin dose was an AUC of 7.5. Since then, multiple large cooperative trials have been performed using AUCs of 6.0 and even 5.0. The lower dosage of carboplatin does not appear to compromise the efficacy of the drugs, and is associated with less toxicity.41-43 Where AUC is as stated above and GFR is the calculated renal function according to the method of Cockcroft and Gault: GFR (ml/min) = 0.85 x {(140-age)/Scr)} x {wt(kg)/72}.

Where Scr is the serum creatinine level. Investigators will use GFR of 125ml/min as cutoff as per NCI guidelines.

Following 6 cycles of IV/IP chemotherapy, a CT of chest, abdomen and pelvis should be obtained for disease surveillance prior to proceeding with radiotherapy (See section 5.4). If clinically indicated, the primary oncologist may have the option to proceed with the CT imaging after 3 cycles of chemotherapy.

5.1.2 Antiemetic Regimens

Nausea and vomiting is anticipated as a side effect. The following representative antiemetic regimen is suggested:

Ondansetron 8-32 mg IV or PO 30 minutes prior to administration of chemotherapy and dexamethasone 10-20 mg IV or PO 30 minutes prior to drug administration.

Aprepitant 125 mg PO one hour prior to chemotherapy on day 1 and 80 mg daily PO on days 2 & 3 for patients having nausea or vomiting with carboplatin (the intravenous formulations may be substituted when available).

Granisetron 10 mcg/kg IV (or 2mg PO) 30 minutes prior to chemotherapy, dexamethasone 10-20 mg IV 30 minutes prior to chemotherapy 5.2 Intraperitoneal device specifications: Insertion of peritoneal catheter may be done by the following procedures as listed below: 1) at time of original laparotomy 2) laparoscopic placement 3) interventional radiology guided placement. Silicone catheters are preferred. Controversy exists between the use of venous 9.6 silicone catheters or silicone IP ports with fenestrations. Bardport silicone peritoneal catheter 14.3 Fr (Reorder number 0603006) is the preferred catheter. This has been FDA approved for IP therapy. The 9.6 Fr single lumen IV access device is also acceptable. Equivalent or similar devices are acceptable if silicone large enough not to kink and without a Dacron cuff.

Procedure at time of original laparotomy:

1. AT the completion of the laparotomy just prior to closing the incision, make a 3-4 centimeter incision over the lower costal margin on the side where the catheter is to be placed. The incision is carried down to the fascia using blunt and sharp dissection.
2. A subcutaneous pocket superior to the incision is fashioned slightly larger than the diameter of the portal.
3. Select an area several centimeters below and lateral to the umbilicus as the peritoneal entrance site of the catheter. Prepare a subcutaneous tunnel from the portal pocket to the site in the peritoneal cavity for the catheter to enter the abdomen and draw the catheter through the subcutaneous tissue into the abdomen using a tunneling device.
4. Attach the catheter to the portal as per manufacturer's instructions and suture the portal in place with permanent suture (i.e. 2-0 prolene) to the fascia overlying the rib cage. Be sure the chemotherapy nurses will be able to feel the port and stabilize it on the chest wall for easy access with Huber needle in the future. Be sure the Huber needle will not have to go through the wound to access the port; the port should lie superior to the port incision site.
5. After flushing the system with heparin 100 units per ml to determine that flow is not obstructed and no leaks exist, place the distal end of the catheter to the desired infusion site, with at least 10 cm of free catheter in the abdomen. Do not allow the catheter to be long enough to reach the bladder, vagina or rectum.
6. Close incisions and place a Huber needle trans-dermally into the portal if the catheter is going to be irrigated in the immediate postoperative period. Wait a minimum of 24 hours prior to treating patient after IP port placement, and wait for return of gastrointestinal function (regular diet tolerated and normal bowel movement) after major laparotomy.

Postoperative procedure with mini laparotomy (video available at SGO.org and GOG.org)

1. Select a site several centimeters below and lateral to the umbilicus and make an incision through skin, subcutaneous tissue and fascia. Separate rectus muscle and enter peritoneum. Knowledge of the previous surgical resections and current anatomy will assist in choosing location.
2. Pull the catheter from subcutaneous tissue into the peritoneal cavity through the full thickness of the abdominal wall (fascia, muscle, peritoneum) from an adjacent location (not through the incision) while under direct visualization to prevent injury to bowel. This can be accomplished with a tonsil clamp or tunneling device.
3. The catheter must be left in the abdominal cavity at least 10 cm to prevent migration out of the peritoneal cavity.
4. The opposite end of the catheter is tunneled up to the costal margin where it is attached to an implanted port as described above. The catheter is left long enough to not retract, but not long enough to reach vagina, rectum or bladder. It is generally left at least 10 cm into the peritoneal cavity.

Post-operative laparoscopically assisted surgical implantation of Port

1. Laparoscopic placement of an IP catheter is usually feasible from a left upper quadrant approach. Knowledge of the previous procedures performed (i.e. bowel resections and anastomosis sites) and location of the tumor will inform the surgeon as to the best approach and what locations to avoid.
2. Once the peritoneal cavity can be visualized, a second puncture can be used to gain access to the peritoneal cavity and then the catheter is tunneled in the subcutaneous tissues to the planned Port pocket.

Port placement under Interventional Radiologic guidance

Interventional radiology may also place IP catheters, if preferred by treating provider. Knowledge of anatomy and the best sites for placement should be communicated between the primary provider or surgeon and the radiologist. CT or ultrasound can allow direct access to peritoneal cavity, followed by subcutaneous tunneling to the anterior chest wall for appropriate port placement and catheter attachment.

Radiation:

Radiation therapy will be delivered at provider discretion after the 6th cycle of chemotherapy.

Physical Factors: All treatment will be delivered by megavoltage equipment ranging from 6 MV to a maximum of 25 MV photons. Cobalt-60 equipment will not be acceptable for treatment on this protocol. Tomotherapy is allowed.

Localization and Simulation Methods: Localization images taken on the conventional or CT-simulator will be necessary in all cases.

Treatment Plan and Dose Specification: Patients may be treated with either conventional radiation therapy approaches or with IMRT. The use of individualized custom blocking is required.

Daily Tumor Dose, Total Dose, and Overall Treatment Time: A daily tumor dose of 180 cGy per day will be given to a total dose of 4500 cGy (180 cGy x 25 treatments) in approximately five weeks. Treatment will be given 5 days a week, from Monday through Friday Dose Distribution (Site): Dose to the CTV should not vary by more than +/- 5% from the prescribed dosage for 3D conformal plans. The use of tissue wedges and/or compensating filters may be necessary to accomplish this goal. As a general rule, only pelvic radiation therapy will be given, unless there is imaging, intra-operative, histologic, or other evidence of para-aortic node involvement.

If there is tumor extension into the vagina, the external beam fields will be modified to include the disease volume with at least a 2 cm margin. For involvement of the distal 1/3 of the vagina, inguino-femoral nodes should also be covered in the external beam RT ports. If the patient's tumor extends into the cervix, or invades deeply and extends into the lower uterine segment, or if there is lymph-vascular space invasion by tumor, or if the tumor has extended into the vagina, such a patient will receive intravaginal boost brachytherapy

Radiation Therapy Volumes and Technique

Pelvic field: 3D Conformal

Portal and Treatment Volume Definition:

The boundaries are as follows:

AP/PA Fields: Cephalad Border:

A transverse line drawn within 2 cm of the L5-S1 interspace or higher if necessary to include known areas of lymph node involvement by tumor.

AP/PA Fields: Caudal Border:

The mid-portion of the obturator foramen or a minimum of 4 cm margin on the vaginal cuff, preferably defined by marker seed placement or by placement of a vaginal swab at the time of simulation.

Lateral Borders: >1 cm beyond the lateral margin of the true pelvis at its widest points.

Alternatively, use of a CT scan to outline the target vessels with a border of at least 1 cm is acceptable.

Lateral Pelvic Fields:

The cephalad and caudal borders are same as above.

Anterior Border:

A horizontal line drawn anterior to the symphysis pubis. When extended in the cephalad direction, this line should pass at least 1 cm anterior to known nodal regions or, in the absence or radiographic documentation, the line should pass at least 1.5 cm anterior to the L5 vertebral body. Individualized custom blocks can be used to achieve this goal.

Posterior Border:

A cephalo-caudal line passing through the third sacral vertebra. Every effort should be made to include the upper vaginal stump with a margin of at least 3 cm.

IMRT Patient Immobilization: Prior to simulation, it is recommended that radiopaque marker be inserted into the vaginal apex to help to identify the area by CT scan. Patients are to be immobilized in the supine position in an immobilization device. Patients are to be treated in the immobilization device. CT scan thickness should be 3 mm or smaller through the region that contains the PTV, extending from at least L3-4 level to below the perineum.

Simulation: CT simulation is required to define clinical target volume (CTV) and planning target volume (PTV). The CT scan should be acquired in the same position and immobilization device as for treatment. The use of IV contrast and bowel prep-contrast are highly recommended for better delineation of the contrast-enhanced pelvic vessels used as a surrogate for regional nodal delineation, as well as small bowel contouring, respectively.

Contouring the Target volumes:

Please refer to the RTOG Gynecological Atlas for volume specification. The atlas may be accessed on the RTOG website at: http://www.rtog.org/gynatlas/main.html The Clinical Target Volume (CTV) is defined as the vaginal apex in addition to pelvic nodal regions lying within the field borders given in Section 4.61. If gas/stool distends the rectum, the CTV is to be expanded to include the anterior half of the rectum to account for evacuation of the rectum. The nodal portion of the CTV should include the internal (hypogastric and obturator), and external iliac lymph node regions. The CTV should be delineated using the contrast enhanced (preferably IV contrast administered) iliac vessels, in addition to the perinodal soft tissue (minimum of 6 mm axial margin around the vessels). Bone and intraperitoneal small bowel should be excluded from the CTV as much as possible (leaving at least 6 mm margin around the vessels). Approximately 1-2 cm of tissue anterior to the sacrum (S1-S3) may be added to the CTV for adequate coverage of pre-sacral nodes, although this is optional and at the discretion of the treating radiation oncologist. In addition the most antero-lateral margin of the external iliac nodes that lie just proximal to the inguinal canal should be excluded from the CTV (nodal CTV should stop at the femoral head). Proximally, the CTV should end 7 mm from the L5-S1 interspace to account for the PTV. The CTV should include the inguino-femoral nodes if the distal one-third of the vagina is involved with tumor.

The PTV should provide a 7 mm-1 cm margin in all directions around the CTV. The definitions of volumes will be in accordance with the 1993 ICRU report #50. Prescribing, recording and reporting photon beam therapy and 1999 ICRU report #62.

Critical normal surrounding structures:

Bladder will be contoured in each slice in which it appears. Rectum will be contoured in each slice in which it appears. As a general guideline, the radiation oncologist can consider the maximum caudal extent of the rectum to lie 1.5-2.0 cm from the bottom of the ischial tuberosities. Superiorly, judgment will be required to establish where the rectum ends and the sigmoid colon begins. The transition to the sigmoid colon is marked by increased curvature and tortuosity in its path. Bowel will be contoured in each slice in which it appears, 2 cm above the PTV as bowel bag and inferiorly to the rectosigmoid junction.

Femoral heads will be contoured in all the slices in which they appear. Constraints: Participants are strongly encouraged to respect the following limits, whether 3-D conformal or IMRT approaches are used.

Small bowel: <30% to receive ≥ 40Gy, Dmax <46 Gy Rectum: < 80% to receive ≥ 40Gy, Dmax <55 Gy Bladder: < 50% to receive ≥ 45Gy, Dmax <60 Gy Femoral heads: < 50% to receive ≥ 40Gy, Dmax <50 Gy.

Radiotherapy

Brachytherapy: If a vaginal brachytherapy boost is to be given based on the criteria given in the protocol. It should commence within 2 weeks of completion of the external beam RT. It should be delivered with a vaginal cylinder (HDR or LDR) or colpostats (LDR), and in the absence of gross residual disease following surgery the treating physician must choose one of the following:

A) HDR: 600 cGy x 2-3, weekly, prescribed at the vaginal surface. Dose optimization should be used in an effort to create reasonable homogeneity of dose around the surface of the applicator. A minimum of 4 cm of vaginal length should be treated.

B) LDR 2000-3500 cGy prescribed at the vaginal surface in 1 insertion at a dose rate of 40-100 cGy/hr. A minimum of 4 cm of vaginal length should be treated.

Physical Factors If an intravaginal boost is to be used, it should be delivered with an intravaginal cylinder (HDR or LDR). Acceptable isotopes include cobalt or iridium for HDR, radium or cesium for LDR.

8.1 Duration of Follow Up Patients will be followed for every 3 months for the first two years, and every 6 months for three years and yearly thereafter, or until death, whichever occurs first. In total, patients will be followed for a maximum of 10 years. Testing such as CA-125 or CT scans may be performed at discretion of the primary physician once off-study. Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event.

10.1 Pre Study Evaluation This evaluation requires completion within 21 days of registration, unless otherwise described. Baseline requirements will consist of a thorough history and physical examination. An ECG < 6 months prior to registration and laboratory tests will be obtained. Tests include, CBC with differential, platelet count, serum chemistry, including electrolytes, creatinine, BUN, glucose, magnesium, calcium, albumin, phosphorous, liver function tests, CA-125, and urinalysis.

Histological documentation of UPSC is required. Pre-study CA125, CT scan of chest, abdomen and pelvis, and CXR (not required if CT of the chest is available) will be obtained.

10.2 Tests during Treatment: Please refer to Appendix A (Study Schedule) Weekly: CBC with differential and platelet count Every 3 weeks (each cycle): CBC with differential and platelet count electrolytes, BUN, creatinine, glucose, magnesium, calcium, phosphorous, albumin, CA125. Every 3 weeks (each cycle): Complete review of systems and complete physical examination, including pelvic examination, clinical evaluation for ototoxicity and neuropathy. Weight and performance status will be documented.

10.3 End of Study Evaluation This evaluation includes a complete history and physical examination and documentation of weight and performance status. Laboratory tests include a complete blood count with differential and platelet count, electrolytes, BUN, creatinine, glucose, magnesium, calcium, phosphorous, albumin, CA125 and urinalysis. CT scan of chest, abdomen and pelvis will be obtained at the completion of the entire IP/carboplatin protocol or earlier if indicated.

10.4 Follow-up Patients will be evaluated every 3 months for the first 2 years and every 6 months for the next 3 years. Evaluation at each visit includes a complete history and physical examination and documentation of weight and performance status. Laboratory tests to be performed in this follow-up period is up to primary provider's discretion, but generally include a complete blood count with differential and platelet count, electrolytes, BUN, creatinine, glucose, magnesium, calcium, phosphorous, albumin, CA125, urinalysis. Surveillance imaging such as CT scan is performed up to provider's discretion, but generally performed annually or earlier if clinically indicated. After a total of 5 years, patients will be seen annually.

ELIGIBILITY:
Inclusion Criteria:

1. Histological/cytologically documented primary FIGO Stage IIIA, IIIB, IIIC1, IIIC2, IVA and IVB uterine serous carcinoma. Patients with stage IVB disease include abdominal sites of metastasis only.
2. All patients must have a procedure for determining the definitive diagnosis of USC. At the discretion of the surgeon, complete surgical staging should include: total hysterectomy, bilateral salpingo-oophorectomy, peritoneal washings, omental biopsy and lymph node evaluation.
3. Residual disease at completion of surgery of ≤ 1cm by surgeon report.
4. Age > 18 years.
5. ECOG performance status of ≤ 2.
6. Written voluntary informed consent.

Exclusion Criteria:

1. Distant metastasis outside the abdominal cavity.
2. Patient has impairment of hepatic, renal or hematologic function as defined by the following baseline laboratory values:

   1. Serum SGOT and /or SGPT > 2.5 times the institutional upper limit of normal (ULN)
   2. Total serum bilirubin > 1.5 mg/dl
   3. Serum creatinine > 2.0 mg/dl
   4. Platelets < 100,000/mm3
   5. Absolute neutrophil count (ANC) < 1500/mm3
   6. Hemoglobin < 8.0 g/dl (the patient may be transfused prior to study entry)
3. History of abdominal/pelvic radiation therapy.
4. Severe or uncontrolled, concurrent medical disease (e.g. uncontrolled diabetes, unstable angina, myocardial infarction within 6 months, congestive heart failure, etc.)
5. Patients with dementia or altered mental status that would prohibit the giving and understanding of informed consent at the time of study entry

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | 2 years post diagnosis
  Number of patients with treatment-related adverse events as assessed by CTCAE v4.0
Feasibility of above regimen in women with advanced stage USC | 2 years post diagnosis
  Feasibility will be assessed by: Treatment completion proportion - the proportion of participants who complete the IV paclitaxel/IP carboplatin followed by IP paclitaxel/RT regimen Screening ratio - the number of potential participants screened per enrolled participant

SECONDARY OUTCOMES:
Patient quality of life | Baseline (after surgery, prior to initiating first cycle), Completion of chemotherapy (18 weeks after Cycle 1 Day 1),Completion of radiation therapy (26 weeks after Cycle 1 Day), Two years post diagnosis
  The questionnaires used are EORTC QLQ-C30. QOL will be assessed using the validated European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-c30) version 3.0. To date, more than 2200 studies using QLQ-C30 have been registered. This 30-item summary score captures the dimension of physical well-being, functional well-being, and symptom scales.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Shih, MD, Principal Investigator — Northwell Health
Locations (1):
- Arisa Kapedani, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sherman ME, Devesa SS. Analysis of racial differences in incidence, survival, and mortality for malignant tumors of the uterine corpus. Cancer. 2003 Jul 1;98(1):176-86. doi: 10.1002/cncr.11484. PMID 12833470
- [Background] Elliott P, Green D, Coates A, Krieger M, Russell P, Coppleson M, Solomon J, Tattersall M. The efficacy of postoperative vaginal irradiation in preventing vaginal recurrence in endometrial cancer. Int J Gynecol Cancer. 1994 Mar;4(2):84-93. doi: 10.1046/j.1525-1438.1994.04020084.x. PMID 11578390
- [Background] Sutton G, Axelrod JH, Bundy BN, Roy T, Homesley H, Lee RB, Gehrig PA, Zaino R. Adjuvant whole abdominal irradiation in clinical stages I and II papillary serous or clear cell carcinoma of the endometrium: a phase II study of the Gynecologic Oncology Group. Gynecol Oncol. 2006 Feb;100(2):349-54. doi: 10.1016/j.ygyno.2005.08.037. Epub 2005 Oct 5. PMID 16213007
- [Result] Abeler VM, Vergote IB, Kjorstad KE, Trope CG. Clear cell carcinoma of the endometrium. Prognosis and metastatic pattern. Cancer. 1996 Oct 15;78(8):1740-7. doi: 10.1002/(sici)1097-0142(19961015)78:83.0.co;2-y. PMID 8859187
- [Result] Gupta D, Gunter MJ, Yang K, Lee S, Zuckerwise L, Chen LM, Goldberg GL, Huang GS. Performance of serum CA125 as a prognostic biomarker in patients with uterine papillary serous carcinoma. Int J Gynecol Cancer. 2011 Apr;21(3):529-34. doi: 10.1097/IGC.0b013e31821091b5. PMID 21436701
- [Result] Major FJ, Blessing JA, Silverberg SG, Morrow CP, Creasman WT, Currie JL, Yordan E, Brady MF. Prognostic factors in early-stage uterine sarcoma. A Gynecologic Oncology Group study. Cancer. 1993 Feb 15;71(4 Suppl):1702-9. doi: 10.1002/cncr.2820710440. PMID 8381710
- [Result] Goff BA, Kato D, Schmidt RA, Ek M, Ferry JA, Muntz HG, Cain JM, Tamimi HK, Figge DC, Greer BE. Uterine papillary serous carcinoma: patterns of metastatic spread. Gynecol Oncol. 1994 Sep;54(3):264-8. doi: 10.1006/gyno.1994.1208. PMID 8088602
- [Result] Hendrickson M, Ross J, Eifel P, Martinez A, Kempson R. Uterine papillary serous carcinoma: a highly malignant form of endometrial adenocarcinoma. Am J Surg Pathol. 1982 Mar;6(2):93-108. doi: 10.1097/00000478-198203000-00002. PMID 7102898
- [Result] Kato DT, Ferry JA, Goodman A, Sullinger J, Scully RE, Goff BA, Fuller AF Jr, Rice LW. Uterine papillary serous carcinoma (UPSC): a clinicopathologic study of 30 cases. Gynecol Oncol. 1995 Dec;59(3):384-9. doi: 10.1006/gyno.1995.9957. PMID 8522260
- [Result] O'Hanlan KA, Levine PA, Harbatkin D, Feiner C, Goldberg GL, Jones JG, Rodriguez-Rodriguez L. Virulence of papillary endometrial carcinoma. Gynecol Oncol. 1990 Apr;37(1):112-9. doi: 10.1016/0090-8258(90)90318-f. PMID 2323606
- [Result] Aalders J, Abeler V, Kolstad P, Onsrud M. Postoperative external irradiation and prognostic parameters in stage I endometrial carcinoma: clinical and histopathologic study of 540 patients. Obstet Gynecol. 1980 Oct;56(4):419-27. PMID 6999399
- [Result] Calais G, Vitu L, Descamps P, Body G, Reynaud-Bougnoux A, Lansac J, Bougnoux P, Le Floch O. Preoperative or postoperative brachytherapy for patients with endometrial carcinoma stage I and II. Int J Radiat Oncol Biol Phys. 1990 Sep;19(3):523-7. doi: 10.1016/0360-3016(90)90476-z. PMID 2211199
- [Result] Carey MS, O'Connell GJ, Johanson CR, Goodyear MD, Murphy KJ, Daya DM, Schepansky A, Peloquin A, Lumsden BJ. Good outcome associated with a standardized treatment protocol using selective postoperative radiation in patients with clinical stage I adenocarcinoma of the endometrium. Gynecol Oncol. 1995 May;57(2):138-44. doi: 10.1006/gyno.1995.1115. PMID 7729725
- [Result] Greven KM, Curran WJ Jr, Whittington R, Fanning J, Randall ME, Wilder J, Peters AJ. Analysis of failure patterns in stage III endometrial carcinoma and therapeutic implications. Int J Radiat Oncol Biol Phys. 1989 Jul;17(1):35-9. doi: 10.1016/0360-3016(89)90367-2. PMID 2745205
- [Result] Greven KM, Lanciano RM, Corn B, Case D, Randall ME. Pathologic stage III endometrial carcinoma. Prognostic factors and patterns of recurrence. Cancer. 1993 Jun 1;71(11):3697-702. doi: 10.1002/1097-0142(19930601)71:113.0.co;2-u. PMID 8490920
- [Result] Greven KM, Randall M, Fanning J, Bahktar M, Duray P, Peters A, Curran WJ Jr. Patterns of failure in patients with stage I, grade 3 carcinoma of the endometrium. Int J Radiat Oncol Biol Phys. 1990 Sep;19(3):529-34. doi: 10.1016/0360-3016(90)90477-2. PMID 2211200
- [Result] Grigsby PW, Perez CA, Camel HM, Kao MS, Galakatos AE. Stage II carcinoma of the endometrium: results of therapy and prognostic factors. Int J Radiat Oncol Biol Phys. 1985 Nov;11(11):1915-23. doi: 10.1016/0360-3016(85)90272-x. PMID 4055452
- [Result] Lanciano RM, Curran WJ Jr, Greven KM, Fanning J, Stafford P, Randall ME, Hanks GE. Influence of grade, histologic subtype, and timing of radiotherapy on outcome among patients with stage II carcinoma of the endometrium. Gynecol Oncol. 1990 Dec;39(3):368-73. doi: 10.1016/0090-8258(90)90268-p. PMID 2258085
- [Result] Mayr NA, Wen BC, Benda JA, Sorosky JI, Davis CS, Fuller RW, Hussey DH. Postoperative radiation therapy in clinical stage I endometrial cancer: corpus, cervical, and lower uterine segment involvement--patterns of failure. Radiology. 1995 Aug;196(2):323-8. doi: 10.1148/radiology.196.2.7617840.
- [Result] Morrow CP, Bundy BN, Kurman RJ, Creasman WT, Heller P, Homesley HD, Graham JE. Relationship between surgical-pathological risk factors and outcome in clinical stage I and II carcinoma of the endometrium: a Gynecologic Oncology Group study. Gynecol Oncol. 1991 Jan;40(1):55-65. doi: 10.1016/0090-8258(91)90086-k. PMID 1989916
- [Result] Randall ME, Wilder J, Greven K, Raben M. Role of intracavitary cuff boost after adjuvant external irradiation in early endometrial carcinoma. Int J Radiat Oncol Biol Phys. 1990 Jul;19(1):49-54. doi: 10.1016/0360-3016(90)90133-5. PMID 2380095
- [Result] Sutton G, Axelrod JH, Bundy BN, Roy T, Homesley HD, Malfetano JH, Mychalczak BR, King ME. Whole abdominal radiotherapy in the adjuvant treatment of patients with stage III and IV endometrial cancer: a gynecologic oncology group study. Gynecol Oncol. 2005 Jun;97(3):755-63. doi: 10.1016/j.ygyno.2005.03.011. PMID 15913742
- [Result] Mackillop WJ, Pringle JF. Stage III endometrial carcinoma. A review of 90 cases. Cancer. 1985 Nov 15;56(10):2519-23. doi: 10.1002/1097-0142(19851115)56:103.0.co;2-m. PMID 2412690
- [Result] Martinez A, Podratz K, Schray M, Malkasian G. Results of whole abdominopelvic irradiation with nodal boost for patients with endometrial cancer at high risk of failure in the peritoneal cavity. A prospective clinical trial at the Mayo Clinic. Hematol Oncol Clin North Am. 1988 Sep;2(3):431-46. PMID 3053592
- [Result] Smith RS, Kapp DS, Chen Q, Teng NN. Treatment of high-risk uterine cancer with whole abdominopelvic radiation therapy. Int J Radiat Oncol Biol Phys. 2000 Oct 1;48(3):767-78. doi: 10.1016/s0360-3016(00)00724-0. PMID 11020574
- [Result] Randall ME, Filiaci VL, Muss H, Spirtos NM, Mannel RS, Fowler J, Thigpen JT, Benda JA; Gynecologic Oncology Group Study. Randomized phase III trial of whole-abdominal irradiation versus doxorubicin and cisplatin chemotherapy in advanced endometrial carcinoma: a Gynecologic Oncology Group Study. J Clin Oncol. 2006 Jan 1;24(1):36-44. doi: 10.1200/JCO.2004.00.7617. Epub 2005 Dec 5. PMID 16330675
- [Result] Thigpen JT, Brady MF, Homesley HD, Malfetano J, DuBeshter B, Burger RA, Liao S. Phase III trial of doxorubicin with or without cisplatin in advanced endometrial carcinoma: a gynecologic oncology group study. J Clin Oncol. 2004 Oct 1;22(19):3902-8. doi: 10.1200/JCO.2004.02.088. PMID 15459211
- [Result] Ball HG, Blessing JA, Lentz SS, Mutch DG. A phase II trial of paclitaxel in patients with advanced or recurrent adenocarcinoma of the endometrium: a Gynecologic Oncology Group study. Gynecol Oncol. 1996 Aug;62(2):278-81. doi: 10.1006/gyno.1996.0227. PMID 8751561
- [Result] Fleming GF, Brunetto VL, Cella D, Look KY, Reid GC, Munkarah AR, Kline R, Burger RA, Goodman A, Burks RT. Phase III trial of doxorubicin plus cisplatin with or without paclitaxel plus filgrastim in advanced endometrial carcinoma: a Gynecologic Oncology Group Study. J Clin Oncol. 2004 Jun 1;22(11):2159-66. doi: 10.1200/JCO.2004.07.184. PMID 15169803
- [Result] Moore KN, Fader AN. Uterine papillary serous carcinoma. Clin Obstet Gynecol. 2011 Jun;54(2):278-91. doi: 10.1097/GRF.0b013e318218c755. PMID 21508697

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT04030000/Prot_SAP_000.pdf